CLINICAL TRIAL: NCT02285920
Title: Safety and Cardiovascular Efficacy of Spironolactone in Dialysis-Dependent End-Stage Renal Disease (ESRD) (SPin-D) Trial
Brief Title: Safety and Cardiovascular Efficacy of Spironolactone in Dialysis-Dependent ESRD Trial
Acronym: SPin-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Brigham and Women's Hospital (Other); George Washington University (Other); Vanderbilt University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 821193
Record Dates: First submitted 2014-10-13; First posted 2014-11-07 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: End-Stage Renal Disease
Keywords: hemodialysis; spironolactone; cardiac fibrosis; diastolic function
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Spironolactone 12.5 mg (Active Comparator): Participants will initiate treatment at 12.5 mg daily and continue at this dose for 36 weeks.
  Interventions: Drug: Spironolactone
- Spironolactone 25 mg (Active Comparator): Participants will initiate treatment at 12.5 mg daily for 2 weeks at which time the dose will be increased to 25 mg daily for a total treatment time of 36 weeks.
  Interventions: Drug: Spironolactone
- Spironolactone 50 mg (Active Comparator): Participants will initiate treatment at 12.5 mg daily for 2 weeks at which time the dose will be increased to 25 mg daily for 2 weeks, and increased to 50 mg daily for a total treatment time of 36 weeks.
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Participants will be treated with placebo for 36 weeks.
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — The trial will be conducted in 2 phases - a dose escalation phase (6 weeks) and a treatment phase (30 weeks). At the end of the dose escalation phase, participants will continue treatment based on the randomized dose assignment for an additional 30 weeks (treatment phase) such that the total duration of study medication is 36 weeks.

SUMMARY:
The SPin-D Trial is a phase II randomized, double-blind, placebo-controlled, multi-center study of spironolactone (SPL) for patients with hemodialysis-dependent end-stage renal disease.

DETAILED DESCRIPTION:
The primary objective of this study is to characterize the safety and tolerability of multiple doses of chronic SPL therapy compared with placebo in maintenance hemodialysis patients and to assess the feasibility of conducting a full-scale, mortality-powered trial of SPL. The effects of SPL compared with placebo on multiple cardiovascular efficacy parameters will also be analyzed. The primary efficacy parameter will be the change in the E' measurement on tissue Doppler echocardiography (TDI) as an index of diastolic function and a surrogate for myocardial fibrosis. Secondary cardiac parameters of interest that will be studied in the overall population or in sub-studies include heart rate variability, circulating markers of fibrosis, and coronary flow reserve (CFR) as an index of microvascular function. These parameters are designed to broaden insight into the potential effects of SPL on cardiac structure and function in individuals with dialysis-dependent ESRD and to assess the feasibility of conducting a full-scale, mortality-powered trial.

ELIGIBILITY:
Inclusion Criteria:

1. Maintenance hemodialysis therapy for end-stage renal disease
2. Age 18-85 years
3. ≥3 calendar months since dialysis initiation. Note if a patient has been on dialysis for ≥3 but less than 6 calendar months, there must be no hospitalizations during the 6 weeks prior to screening, and no change in estimated dry weight (EDW) within 2 weeks of the screening date.
4. For women of childbearing potential, willingness to use a highly effective method of birth control for up to 4 weeks after the last dose to study drug.
5. Ability to provide informed consent

Exclusion Criteria:

1. Serum potassium ≥6.5 mEq/L within the 3 months prior to screening
2. Serum potassium level ≥6.0 mEq/L within 2 weeks prior to the baseline visit. If a potassium value is not available through routine clinical care during this 2-week period a potassium measurement will be performed as a research test.
3. Unscheduled dialysis for hyperkalemia within the 3 months prior to screening
4. Pre-dialysis systolic blood pressure <100 mm Hg within 2 weeks prior to screening or at the baseline visit
5. 2 or more dialysis sessions within the month prior to screening with either 2 intra-dialytic measurements of systolic blood pressure <80 mm Hg or muscle cramping, light-headedness, nausea or hypotension requiring infusion of saline or other intervention directed at hypotension
6. Current dual use of angiotensin converting enzyme inhibitor (ACEI) and angiotensin receptor blocker (ARB)
7. Current use of digoxin
8. Current use of spironolactone or eplerenone
9. Allergy to spironolactone
10. Inability to maintain dialysis machine blood flow ≥300 mL/min during any of the most recent 3 dialysis sessions prior to the screening visit as an indicator of vascular access dysfunction
11. Mitral valve repair or replacement
12. Severe mitral valve disease by echocardiography, coronary angiography or cardiac magnetic resonance imaging
13. Anticipated kidney transplant, change to peritoneal dialysis, or transfer to another dialysis unit within 9 months
14. Expected survival <9 months
15. Pregnancy, anticipated pregnancy, or breastfeeding
16. Incarceration
17. Participation in another intervention study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-11; Primary Completion 2017-06 (Actual); Study Completion 2017-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Dember, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - The George Washington University, Washington D.C., District of Columbia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Kidney Research Institute, University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Started | 51 | 27 | 26 | 25
Completed | 47 | 23 | 21 | 24
Not Completed | 4 | 4 | 5 | 1
Not completed — Kidney transplantation | 2 | 2 | 2 | 0
Not completed — Change to peritoneal dialysis | 0 | 0 | 1 | 0
Not completed — Transfer to non-participating unit | 0 | 1 | 0 | 0
Not completed — Dialysis discontinuation | 0 | 1 | 0 | 0
Not completed — Death | 2 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Participants were enrolled from dialysis units affiliated with four U.S. academic medical centers. The Institutional Review Boards affiliated with the clinical centers and with the data coordinating center approved the protocol and all participants provided informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg | Total
Number analyzed (Participants) | 51 | 27 | 26 | 25 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (11.5) | 55.1 (13.6) | 53.3 (13.5) | 55.5 (9.8) | 55.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 7 | 6 | 44
  Male | 32 | 15 | 19 | 19 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 2 | 2 | 11
  Not Hispanic or Latino | 47 | 24 | 24 | 23 | 118
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 39 | 18 | 18 | 17 | 92
  White | 7 | 8 | 7 | 5 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety - Number of Participants With Serum Potassium >6.5 mEq/L
Description: The number of participants who had serum potassium >6.5 mEq/L was assessed by treatment arm.
Time Frame: 0 - 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 51 | 27 | 26 | 25
Participants | 9 | 4 | 4 | 8

2. Primary Outcome: Safety - Participants With Serious Hypotension
Description: The number of participants experiencing serious hypotension, defined as hypotension requiring hospitalization or ED visit and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection).
Time Frame: 0 - 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 51 | 27 | 26 | 25
Participants | 0 | 2 | 0 | 3

3. Primary Outcome: Study Drug Tolerability
Description: Tolerability is defined as number of participants who experienced permanent study drug discontinuation or dose reduction.
Time Frame: 0 - 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 51 | 27 | 26 | 25
Participants | 16 | 5 | 6 | 8

4. Primary Outcome: Efficacy - Change in Mitral Annular E' Velocity
Description: Change in mitral annular E' velocity measured using Tissue Doppler Index (TDI) echocardiography. Efficacy outcomes were considered exploratory with a goal of detecting signals rather than clearly demonstrating efficacy.
Time Frame: Baseline to 36 weeks
Population: The number of participants analyzed reflects those who had analyzable echocardiogram data at both study time points.
Measure: Mean (Standard Deviation); unit: cm/second
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 40 | 20 | 15 | 22
cm/second
  Baseline MA E' | 7.4 (1.7) | 7.6 (1.8) | 7.8 (1.9) | 7.0 (1.9)
  36 Week MA E' | 7.5 (1.9) | 7.4 (1.9) | 7.7 (1.4) | 7.3 (1.9)
  Change between baseline - 36 weeks | 0.1 (1.1) | -0.2 (1.0) | -0.1 (1.2) | 0.3 (1.6)

5. Primary Outcome: Feasibility of Conducting a Full-scale Mortality-powered Trial
Description: An objective of this study is to assess the feasibility of conducting a full-scale mortality-powered trial. Feasibility assessed based on recruitment, dropout and loss to follow-up rates.
Time Frame: 0 - 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 51 | 27 | 26 | 25
Participants
  Kidney transplantation | 2 | 2 | 2 | 0
  Change to peritoneal dialysis | 0 | 0 | 1 | 0
  Transfer to non-participating facility | 0 | 1 | 0 | 0
  Dialysis discontinued | 0 | 1 | 0 | 0
  Death | 2 | 0 | 2 | 1
  Study completed | 47 | 23 | 21 | 24

6. Secondary Outcome: Safety - Number of Participants With Serious Hyperkalemia
Description: Number of patients with serious hyperkalemia requiring hospitalization, emergency/unscheduled dialysis or resin therapy
Time Frame: 0 - 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 51 | 27 | 26 | 25
Participants | 6 | 2 | 0 | 7

7. Secondary Outcome: Safety - Hyperkalemia Requiring Adjustment in Treatment
Description: Hyperkalemia requiring adjustment in dialysate potassium concentration, or discontinuation of study medication
Time Frame: 0 - 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 51 | 27 | 26 | 25
Participants | 13 | 2 | 5 | 7

8. Secondary Outcome: Safety - Inter- or Intra-dialytic Hypotension
Description: Inter- or intra-dialytic hypotension defined as:
  1. Inter-dialytic: systolic blood pressure <90 mm Hg or inter-dialytic hypotension requiring adjustment in anti-hypertensive medications or treatment in a hospital or emergency room.
  2. Intra-dialytic: systolic blood pressure <80 mm Hg during ≥3 dialysis sessions per 30-day period or treatment for either hypotension or symptoms of hypotension during ≥3 dialysis sessions per 30-day period
Time Frame: 0 - 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 51 | 27 | 26 | 25
Participants
  Inter-dialytic hypotension only | 3 | 1 | 1 | 0
  Intra-dialytic hypotension only | 20 | 9 | 8 | 14
  Inter- & intra-dialytic hypotension | 3 | 3 | 5 | 5
  No inter- or intra-dialytic hypotension | 25 | 14 | 12 | 6

9. Secondary Outcome: Safety - Cardiovascular Death
Description: Number of Cardiovascular deaths defined as death due to myocardial infarction, congestive heart failure, cardiac valvular disease, arrhythmia, sudden death, stroke, or peripheral arterial disease
Time Frame: 0 - 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 51 | 27 | 26 | 25
Participants | 1 | 0 | 2 | 1

10. Secondary Outcome: Efficacy - Secondary Cardiac Outcome Measure - Left Ventricular Ejection Fraction (LVEF)
Description: Secondary outcome measures include other echocardiographic markers of systolic and diastolic function
  • Change in left ventricular ejection fraction between Baseline and 36 weeks
Time Frame: Baseline - 36 weeks
Population: The number of participants analyzed reflects those who had analyzable echocardiogram data at both study time points.
Measure: Mean (Standard Deviation); unit: percent ejection fraction
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 48 | 24 | 19 | 24
percent ejection fraction
  LVEF Baseline | 68.9 (4.0) | 65.9 (8.5) | 66.0 (11.4) | 68.2 (5.8)
  LVEF 36-Week | 70.7 (3.1) | 66.9 (9.9) | 65.3 (13.9) | 69.5 (6.3)
  LVEF Change | 1.8 (4.1) | 1.0 (4.7) | -0.7 (7.3) | 1.3 (3.7)

11. Secondary Outcome: Efficacy - Secondary Cardiac Outcome Measures Left Ventricular Mass Index (LVMI)
Description: Secondary outcome measures include other echocardiographic markers of systolic and diastolic function,
  • Change in left ventricular mass index (LVMI) between baseline and 36 weeks
Time Frame: Baseline - 36 weeks
Population: The number of participants analyzed reflects those who had analyzable echocardiogram data at both study time points.
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 48 | 24 | 19 | 24
g/m^2
  LVMI Baseline | 105.2 (25.2) | 115.5 (26.7) | 116.4 (26.9) | 106.3 (29.2)
  LVMI 36-Week | 94.8 (22.4) | 104.6 (27.0) | 109.1 (30.5) | 96.5 (25.7)
  LVMI Change | -10.4 (11.9) | -10.9 (18.1) | -7.3 (21.0) | -9.8 (9.3)

12. Secondary Outcome: Efficacy - Secondary Cardiac Outcome Measures - Ratio of Mitral Peak Velocity to Diastolic Mitral Annular Velocity (E/E')
Description: Secondary outcome measures include other echocardiographic markers of systolic and diastolic function,
  • E/E' is the ratio of mitral peak velocity of early filling (E) to early diastolic mitral annular velocity (E')
Time Frame: Baseline - 36 weeks
Population: The number of participants analyzed reflects those who had analyzable echocardiogram data at both study time points.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 48 | 24 | 19 | 24
ratio
  E/E' Baseline | 10.7 (5.8) | 11.8 (6.2) | 9.2 (5.0) | 12.5 (5.6)
  E/E' 36-Week | 11.5 (7.0) | 12.2 (80.) | 10.6 (3.9) | 11.9 (5.5)
  E/E' Change | 0.9 (3.6) | 0.4 (4.4) | 1.4 (2.2) | -0.6 (4.0)

13. Secondary Outcome: Efficacy - Secondary Cardiac Outcome Measures - Left Ventricular Global Longitudinal Strain (LVGLS)
Description: Secondary outcome measures include other echocardiographic markers of systolic and diastolic function,
  • Change in myocardial strain and strain rate between baseline and 36 weeks
Time Frame: Baseline - 36 weeks
Population: The number of participants analyzed reflects those who had analyzable echocardiogram data at both study time points.
Measure: Mean (Standard Deviation); unit: % of myocardial shortening
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 48 | 24 | 19 | 24
% of myocardial shortening
  LVGLS Baseline | -17.2 (2.8) | -16.7 (3.3) | -17.2 (4.2) | -17.4 (3.0)
  LVGLS 36-week | -18.1 (2.8) | -17.0 (3.3) | -17.0 (3.9) | -18.2 (3.0)
  LVGLS Change | -0.8 (2.3) | -0.3 (3.3) | 0.2 (2.7) | -0.7 (2.9)

14. Secondary Outcome: Safety - Combined Incidence of Potassium >6.5 mEq/L or Serious Hyperkalemia
Description: The number of participants who had serum potassium >6.5 mEq/L or serious hyperkalemia was assessed by treatment arm.
Time Frame: 0 - 40 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
Number analyzed (Participants) | 51 | 27 | 26 | 25
Participants | 13 | 5 | 5 | 10

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at each study visit during Weeks 1 - 40 of trial participation.
Description: Specific signs and symptoms, anticipated in patients treated with spironolactone, were collected on the Adverse Event of Interest form.
  Adverse events are reported according to the MedDRA hierarchy. The System Organ Class is comprised of a variety of related High Level Group Terms.
Arm/Group | Placebo | Spironolactone 12.5 mg | Spironolactone 25 mg | Spironolactone 50 mg
All-Cause Mortality (participants affected / at risk) | 2/51 | 0/27 | 2/26 | 1/25
Serious Adverse Events (participants affected / at risk) | 27/51 | 13/27 | 13/26 | 12/25
Other Adverse Events (participants affected / at risk) | 45/51 | 24/27 | 25/26 | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | Spironolactone 12.5 mg (N=27) | Spironolactone 25 mg (N=26) | Spironolactone 50 mg (N=25)
Anemia (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 2 (3) | 2 (2)
Acute MI, atrial fibrillation, bradycardia, palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Abdominal pain, diarrhea, GI hemorrhage, nausea, vomiting (Gastrointestinal disorders) | 7 (19) | 2 (8) | 5 (8) | 3 (4)
Asthenia, chest pain (General disorders) | 6 (7) | 3 (3) | 6 (10) | 2 (6)
Hemobilia, hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bacteremia, influenza, osteomyelitis, pneumonia. sepsis, skin graft infection, UTI, viral infection (Infections and infestations) | 4 (4) | 1 (2) | 6 (7) | 5 (7)
AVfistula site hemorrhage, vascular access complications, fall, laceration, rib fracture (Injury, poisoning and procedural complications) | 6 (10) | 5 (5) | 5 (5) | 3 (4)
Cardiac catheterisation, fistulogram, pleural biopsy (Investigations) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Hyperkalemia, hypocalcemia, fluid overload (Metabolism and nutrition disorders) | 6 (8) | 3 (4) | 0 (0) | 6 (14)
Arthralgia, back pain, neck pain, extremity pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 1 (1) | 3 (6)
Gastric cancer, renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Balance disorder, dementia, headache, paralysis, syncope (Nervous system disorders) | 3 (4) | 3 (4) | 1 (1) | 0 (0)
Anxiety, depression, mental status changes (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bladder mass, hematuria, urinary retention (Renal and urinary disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Asthma, COPD, cough , dyspnea, pleural effusion, stridor (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 4 (4) | 5 (13) | 3 (3)
Blister, erythema, pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Angioplasty, catheter placement, toe amputation, renal transplant, thrombectomy, nephrectomy (Surgical and medical procedures) | 6 (6) | 3 (4) | 3 (4) | 5 (6)
Hypertension, hypotension, thrombosis (Vascular disorders) | 2 (4) | 5 (6) | 0 (0) | 4 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | Spironolactone 12.5 mg (N=27) | Spironolactone 25 mg (N=26) | Spironolactone 50 mg (N=25)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (6) | 1 (1) | 3 (4)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 4 (8) | 4 (5) | 6 (13) | 6 (11)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain, nausea, diarrhea, constipation (Gastrointestinal disorders) | 12 (23) | 10 (16) | 7 (21) | 6 (7)
Pain, peripheral edema, malaise (General disorders) | 8 (10) | 1 (1) | 3 (3) | 0 (0)
Bronchitis, diverticulitis, cystitis, cellulitis, naspharyngitis (Infections and infestations) | 7 (11) | 4 (5) | 5 (6) | 4 (4)
Fall, rib fracture, vascular graft complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1) | 3 (4)
Skin biopsy, liver biopsy, low hemoglobin (Investigations) | 3 (5) | 3 (3) | 0 (0) | 2 (2)
Hyperkalemia, hyperphosphatemia, hypercalcemia, gout (Metabolism and nutrition disorders) | 22 (70) | 10 (26) | 11 (34) | 10 (39)
Arthralgia, arthritis, osteoarthritis, tendonitis, neck pain (Musculoskeletal and connective tissue disorders) | 6 (12) | 3 (4) | 4 (4) | 4 (10)
Dizziness, headache, migraine, tremor, syncope (Nervous system disorders) | 4 (5) | 2 (2) | 5 (9) | 2 (5)
Dysuria, hematuria, incontinence (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Breast tenderness, enlargement (Reproductive system and breast disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (3)
COPD, pleural effusion, asthma, cough, dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (5) | 2 (3) | 1 (1)
Pruritis, rash (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 1 (1) | 2 (2)
AV fistula, thrombectomy, catheter placement, stent placment, amputation, vascular operation (Surgical and medical procedures) | 3 (7) | 4 (5) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 25 (90) | 14 (30) | 13 (46) | 17 (75)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT02285920/Prot_SAP_000.pdf